CLINICAL TRIAL: NCT00332826
Title: A Phase 3, 12-month Treatment, Multicenter, Randomized, Open-Label, Parallel Group Clinical Trial Comparing Prandial Subcutaneous Insulin With Prandial Inhaled Technosphere Insulin in Subjects With Diabetes Mellitus and Asthma
Brief Title: Inhaled Technosphere Insulin in Subjects With Diabetes Mellitus and Asthma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Non-safety related business decision to combine special population protocols
Sponsor: Mannkind Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-105
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Asthma
Keywords: Inhaled insulin; Diabetes Type I and II with Asthma
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Asthma

INTERVENTIONS:
Drug: Technosphere Insulin

SUMMARY:
The clinical trial is designed to evaluate the safety of inhaled Technosphere/Insulin compared with non-inhaled anti-diabetic therapies in subjects with type 1 or type 2 diabetes mellitus and concurrent asthma.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Step 1 to 3 asthma as per the NAEPP guidelines
* Clinical diagnosis of Type 1 or Type 2 diabetes mellitus for at least 1 year
* Current stable anti-diabetic regimen (insulin alone or in combination with oral anti-hyperglycemic agents)
* Subjects must exhibit <30% variability in PEF measurements during the 2 week run in period.
* Subjects must not meet any criteria for exacerbations of asthma during the 2 week run in period
* Body mass index (BMI) < 40kg/m2
* HbA1c >6.0% to <11.5%

Exclusion Criteria:

* Severe complications of diabetes in the opinion of the investigator
* Seizure disorder
* Significant cardiovascular dysfunction and/or history within 3 months of screening
* Hypertension with systolic blood pressure of !80 mm Hg and/or diastolic blood pressure >110 mm HG at screening despite pharmacologic therapy.
* Clinical nephrotic syndrome or renal dysfunction or disease
* Total daily insulin requirement of >1.4 U/kg body weight
* Clinical diagnosis of Step 4 asthma
* Use of >6 puffs/day of fast acting bronchodilator
* Currently using an insulin delivery pump
* Use of Pramlintide acetate or any incretins must be discontinued 8 weeks prior to screening
* Two or more severe hypoglycemic episodes within the past 6 months.
* Any hospitalization or emergency room visit due to poor diabetic control with 6 months of screening.
* Current use of systemic steroids
* Subjects who currently smoke tobacco or who have smoked within the past 6 months
* Urine cotinine test of > 100ng/ml
* Current drug or alcohol abuse
* Clinically significant abnormalities on screening laboratory evaluation
* Cancer within the past 5 years or any history of lung neoplasms
* History of active and/or cirrhotic hepatic disease and/or abnormal liver enzymes.
* Active infection or history of severe infection with 30 days of screening.
* Anemia
* History of anaphylaxis and/or angioneurotic edema
* Diagnosis of chronic obstructive pulmonary disease (COPE)
* Previous exposure to any inhaled insulin product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The primary safety outcome will be measurements of post bronchodilator FEV1 throughout the treatment period

CONTACTS AND LOCATIONS:
Locations (77):
- United States (25):
  - Arizona Research Center, Phoenix, Arizona
  - Northwest Medical Center, Phoenix, Arizona
  - Premiere Pharmaceutical Research LLC, Tempe, Arizona
  - Canyon Internal Medicine, Tucson, Arizona
  - Associated Pharmaceutical Research Center Inc, Buena Park, California
  - Family Medical Center, Foothill Ranch, California
  - Health Care Partners Medical Group, Long Beach, California
  - Golden Pine Clinical Research, Long Beach, California
  - Keck USC School of Medicine, Los Angeles, California
  - Pinaccle Trials Inc (SMO), Atlanta, Georgia
  - Executive Health and Research Associates Inc, Atlanta, Georgia
  - Atlanta Pharmaceutical Research Center, Dunwoody, Georgia
  - Southeastern Endocrine & Diabetes, Roswell, Georgia
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Franklin Square Hospital, Baltimore, Maryland
  - Healthcare Research, Florissant, Missouri
  - MedEx Healthcare Research Inc(009), St Louis, Missouri
  - Billings Clinic Research Division, Billings, Montana
  - Your Doctors Care, Hillsborough, New Jersey
  - Hopewell Valley Family Medicine PA, Trenton, New Jersey
  - Eastside Comprehensive Medical Center, New York, New York
  - Carolinas Research, Concord, North Carolina
  - Cleveland Clinic Dept of Endocrinology, Cleveland, Ohio
  - Diabetes & Glandular Disease Research Assoc PA, San Antonio, Texas
  - McLennan County Medical Education and Research Foundation, Waco, Texas
- Argentina (2):
  - DIM (Clinica Privada), Buenos Aires
  - Ins De Inv Cardiovascular La Plata, La Plata
- Brazil (7):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Sao Lucas - PUCRS (Fritscher), Porto Alegre
  - Hospital Nossa Senhora da Conceicao, Porto Alegre
  - Ccbr Brasil Centro de Analises e Pesquisas Clinicas Ltda, Rio de Janeiro
  - CPClin-Centro de Pesquisas Clinicas, São Paulo
  - Clinica de Endocrinologia, São Paulo
- Canada (6):
  - Finchlea Medical Group, Brampton, Ontario
  - Courtice Health Centre, Courtice, Ontario
  - Parkwood Hospital, London, Ontario
  - The London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Albany Medical Center, Toronto, Ontario
  - Windsor Professional Research, Windsor, Ontario
- Czechia (5):
  - Surgery of Diabetology, Mělník, CZE
  - Interni oddeleni nemocnice Na Homolce, Prague, CZE
  - Diabetologicka Outpatient Surgery of Diabetology, Slaný, CZE
  - InternÃ- a diabetologickÃ¡ Outpatient, Ostrava, Ostrava
  - I InternÃ- klinika, Ostrava, Ostrava
- Mexico (4):
  - Hospital Angeles Mocel, Mexico City, Mexico City
  - Mexican Institute of Clinical Research, Mexico City, MX
  - Nuevo Sanatorio Durango, Delegacion Cuauhtemoc
  - Hospital Angeles de las Lomas, Huixquilucan
- Poland (6):
  - Klinika Endocrinologii Diabetologii I, Bialystock, POL
  - NZOZ Specjalistyczny Osrodek Internistyczno - Diabetologiczny, Bialystok, POL
  - Dzial Badan Klinicznych Malopoiskie, Krakow, POL
  - III Oddzial Chorob Wewnetrznych Szpital, Krakow, POL
  - Oddzial Chorob Wewnetrznych Wojewodzki, Lodz, Zgierz
  - Oddzial Kliniczny Diabetologii (009) Kliniczny nr 1 im Norberta Barlickiego Uniwersytety Meycznego, Lodz
- Russia (13):
  - NHI Kemerovo Regional Clinical Hospital, Kemerovo, RUS
  - NI Principal Military Clinical Hospital n a academician N.N. Burdenko, Moscow, RUS
  - Moscow State Medico-Stomatological University City Hospital # 23, Moscow, RUS
  - Central Medical Sanitary Unit #122, Saint Petersburg, RUS
  - City Hospital # 2 Endocrinology Department, Saint Petersburg, RUS
  - Smolensk Medical Academy Smolensk Regional Clinical Hospital, Smolensk, RUS
  - Yaroslavl Municipal Health Care Institution Clinical Hospital for Emergency Care na NV Soloviev, Yaroslavl, RUS
  - Federal State Institution Pulmonology Research Institute of Federal Agency of HC&SD, Moscow
  - City Clinical Hospital #64 Center of Applied Clinical Paharmacology Friendship University, Moscow
  - Central Clinical Hospital of Russian Science Academy, Moscow
  - City Clinical Hospital # 61, Moscow
  - Russian Scientific Center of Restoration Medicine & Balneology, Moscow
  - St Petersburg Medical Academy (Ilkovich), Saint Petersburg
- Hospital 2 de Maig, Barcelona, Barcelona, Spain
- Ukraine (4):
  - Donetsk State Medical University, Donetsk, UKR
  - Railway Clinical Hospital on Donetsk Station, Donetsk, UKR
  - Chair Family Med of National Med University, Kiev, UKR
  - Institute of Endocrinology and Metabolism, Kiev, UKR
- United Kingdom (4):
  - Clinical Research Centre The Royal London Hospital, London, GBR
  - Northern General Hospital, Sheffield, GBR
  - Birmingham Heartland Hospital, West Midlands, GBR
  - Addenbrooke's Hospital Department of Medicine, Cambridge